CLINICAL TRIAL: NCT05163366
Title: Oral Morphine Versus Rectal Ketamine in Pain Management During Burns Wound Dressing Changes in Paediatric Population at Mbarara Regional Referral Hospital: An Open Label Randomized Trial
Brief Title: Oral Morphine Versus Ketamine in Pain Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/ANDREW
Record Dates: First submitted 2021-04-22; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-04

CONDITIONS: Pain, Procedural
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Rectal ketamine versus oral morphine in pain management in paediatric wound and burns
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Experimental): Group A will receive rectal ketamine(Ket)
  Interventions: Drug: GROUP A
- GROUP B (Active Comparator): Group B will receive only traditional standard of care protocols.
  Interventions: Drug: GROUP B

INTERVENTIONS:
Drug: GROUP A — Rectal Ketamine will be administered at 6 mg/kg and with a rectal nozzle it's infused through the rectum. The rectal ketamine will be administered after scoring pain just before the start of the procedure and then about 15 minutes later the procedure will start when the patient has achieved a nystagmus.
  Other Names: KETAMINE GROUP
  Arms: GROUP A
Drug: GROUP B — The tradition standard protocols involve the use of 0.3mg/kg of oral morphine about an hour before the start of the procedure before the start of the procedure to allow for the onset of action of oral morphine for every single procedure in this arm.
  Other Names: MORPHINE GROUP
  Arms: GROUP B

SUMMARY:
The study will mainly focus on procedural pain management using oral morphine versus rectal ketamine during paediatric burn and wound dressing at Mbarara Regional Referral Hospital.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to one of the two treatment groups A and B. Guardians of patients who are scheduled for burn wound care will sign written consent pre- operatively about procedural pain management. Group A will receive rectal ketamine while those in Group B will receive only traditional standard of care protocols.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 6 months and 6-years old scheduled for a minimum of one procedure for burn wound dressing at the pediatric unit at Mbarara Regional Referral Hospital

Exclusion Criteria:

* Children with rectal or anal pathology,
* Refusal to assent to participate or parental or guardian refusal to consent in the study
* Children who require mechanical ventilation or already intubated in Intensive care unit
* Those allergic to Ketamine or its constituents

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
PAIN SCORES ON ORAL MORPHINE VERSUS KETAMINE ARM | 4 hours
  The primary endpoint will be difference in pain scores on a Revised FLACC(Face, Leg, Activity, Cry, Consolability) scale in the two arms.The primary endpoint will be difference in pain scores on a Revised FLACC(Face, Leg, Activity, Cry, Consolability) scale in the two arms. Each category is scored on the 0-2 scale, which results in a total score of 0-10. 0: Relaxed and comfortable, 1-3 : Mild discomfort ,4-6 : Moderate pain, 7-10 : Severe discomfort or pain or both
DIFFERENCE IN THE INCIDENCE OF ADVERSE EFFECTS IN ORAL MORPHINE VERSUS KETAMINE ARM | 4 hours
  Secondary endpoint will be the difference in the incidence of adverse effects a cross arms obtained from patient, nurse, and chart for DAIDS Adverse Event Grading Table 2014.

CONTACTS AND LOCATIONS:
Overall Officials: ALICE G. ATAI, MbChB, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, Uganda